CLINICAL TRIAL: NCT03481296
Title: Culturally Adapted Multilevel Decision Support Navigation Trial To Reduce Colorectal Cancer Disparity Among At-Risk Asian American Primary Care Patients
Brief Title: Screening TO Prevent ColoRectal Cancer (STOP CRC) Among At-Risk Chinese and Korean American Primary Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Thomas Jefferson University (Other); University of Maryland, College Park (Other)
Responsible Party: Principal Investigator, Sunmin Lee, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01MD012778 [2020-5953]; 1R01MD012778-01A1 (NIH)
Record Dates: First submitted 2018-03-02; First posted 2018-03-29 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer Screening; Asian Americans; Patient Navigation; Decision Counseling Program
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advanced Control (Active Comparator): The advanced control group receives a set of standard materials regarding colorectal cancer screening.
  Interventions: Behavioral: Advanced Control
- Culturally Adapted Decision Support Navigation Intervention (Experimental): The culturally adapted decision support navigation intervention group receives everything advanced group receives as well as decision support and navigation contacts.
  Interventions: Behavioral: Culturally-Adapted Decision Support Navigation Intervention

INTERVENTIONS:
Behavioral: Advanced Control — Participants receive linguistically and culturally tailored information booklet on colorectal cancer and colorectal cancer screening, colonoscopy instructions, stool blood test kits and reminder by mail. Participants' height, weight, and waist/hip circumference, blood pressure, blood glucose, and cholesterol levels will be measured by trained research staff. Participants will also receive the result of body measurements right away as a free service.
  Arms: Advanced Control
Behavioral: Culturally-Adapted Decision Support Navigation Intervention — Participants in this group receive everything that advanced control group receives. In addition to a set of standard materials, they receive culturally and linguistically adapted decision counseling from the patient navigator. The patient navigator develops an individualized colorectal cancer screening plan using a theory-based online Decision Counseling Program. After the Program is completed, the patient navigator develops individualized colorectal cancer screening plan and shares the information with participants and participants' primary care physicians. Then, primary care physicians encourage the colorectal cancer screening to participants.
  Arms: Culturally Adapted Decision Support Navigation Intervention

SUMMARY:
The objective of the study is to conduct a randomized controlled trial to determine the impact of a multi-level culturally-sensitive decision support intervention on colorectal cancer screening adherence among 400 Chinese and Korean American primary care patients.

DETAILED DESCRIPTION:
This study culturally adapts existing evidence-based decision support navigation intervention and tests its efficacy among 200 Chinese and Korean American men and 200 Chinese and Korean American women aged 50 to 75 eligible for colorectal cancer screening. Participants are recruited from primary care physician clinics. The study is designed to compare colorectal cancer screening outcomes between the decision support navigation intervention and the advanced control. Those randomized to the advanced control group only receives an informational booklet, a stool blood test kit and a reminder by mail. Those randomized to the decision support navigation intervention group receives everything the advanced control group receives as well as decision support and navigation contacts. Investigators in the study develop an individualized screening plan using a theory-based online Decision Counseling Program, share the plan with the participants' primary care physicians, and have primary care physicians to encourage the colorectal cancer screening to participants. Using outcomes data collected by survey and medical record review, this study: (1) determines overall colorectal cancer screening adherence in the culturally adapted decision support navigation intervention vs. the advanced control; (2) measures change in colorectal cancer screening decision stage in the culturally adapted decision support navigation intervention vs. the advanced control; and (3) assesses colorectal cancer screening test-specific (stool blood test vs. colonoscopy) adherence in the culturally adapted decision support navigation intervention vs. the advanced control. Additionally, investigators in the study evaluate intervention reach, effectiveness, adoption, implementation, and maintenance using interview data.

ELIGIBILITY:
Inclusion Criteria:

* Male and female Chinese and Korean American patients aged 50 to 75, who are not up to date for colorectal cancer screening

Exclusion Criteria:

* Those with a family history, previous history of removing polyps, inflammatory bowel disease, or diagnosis of colorectal cancer screening.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Colorectal cancer screening adherence at 6 months by medical record review | 6 months
  Measure overall colorectal cancer screening adherence at 6 months by medical record review.
Colorectal cancer screening adherence at 6 months by self-report | 6 months
  Measure overall colorectal cancer screening adherence at 6 months by self-report during 6-month survey (by phone).
Overall colorectal cancer screening adherence at 12 months by medical record review | 12 months
  Measure overall colorectal cancer screening adherence at 12 months by medical record review.
Overall colorectal cancer screening adherence at 12 months by self-report | 12 months
  Measure overall colorectal cancer screening adherence at 12 months by self-report (by phone interview).
Colorectal cancer screening decision stage at baseline (Stool Blood Test) | Baseline
  Measure colorectal cancer screening decision stage for stool blood test at baseline.
Colorectal cancer screening decision stage at 6-months (Stool Blood Test) | 6 months
  Measure colorectal cancer screening decision stage for stool blood test at 6 months.
Change in colorectal cancer screening decision stage between baseline and 6 months (Stool Blood Test) | Baseline and 6 months
  Measure change in colorectal cancer screening decision stage for stool blood test between baseline and 6 months.
Colorectal cancer screening decision stage at baseline (Colonoscopy) | Baseline
  Measure colorectal cancer screening decision stage for colonoscopy at baseline.
Colorectal cancer screening decision stage at 6 months (Colonoscopy) | 6 months
  Measure colorectal cancer screening decision stage for colonoscopy at 6 months.
Change in colorectal cancer screening decision stage between baseline and 6 months (Colonoscopy) | Baseline and 6 months
  Measure change in colorectal cancer screening decision stage for colonoscopy between baseline and 6 months.
Colorectal cancer screening test-specific adherence at 6 months (Stool Blood Test) | 6 months
  Measure the fraction of participants who undergo a stool blood test at 6 months.
Colorectal cancer screening test-specific adherence at 6 months (Colonoscopy) | 6 months
  Measure the fraction of participants who undergo a colonoscopy at 6 months.
Colorectal cancer screening test-specific adherence at 12 months (Stool Blood Test) | 12 months
  Measure the fraction of participants who undergo a stool blood test at 12 months.
Colorectal cancer screening test-specific adherence at 12 months (Colonoscopy) | 12 months
  Measure the fraction of participants who undergo a colonoscopy at 12 months.

SECONDARY OUTCOMES:
Knowledge about colorectal cancer and colorectal cancer screening (Baseline) | Baseline
  Measure knowledge about colorectal cancer and colorectal cancer screening at baseline.
Knowledge about colorectal cancer and colorectal cancer screening (6 months) | 6 months
  Measure knowledge about colorectal cancer and colorectal cancer screening at 6 months.
Change in knowledge about colorectal cancer and colorectal cancer screening between baseline and 6 months | Baseline and 6 months
  Measure change in knowledge score about colorectal cancer and colorectal cancer screening between baseline and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Sunmin Lee, ScD, Principal Investigator — UC Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morey BN, Shi Y, Ryu S, Redline S, Kawachi I, Park HW, Lee S. Risk of sleep apnea associated with higher blood pressure among Chinese and Korean Americans. Ethn Health. 2024 Apr;29(3):295-308. doi: 10.1080/13557858.2024.2311417. Epub 2024 Feb 2. PMID 38303653
- [Derived] Morey BN, Ryu S, Shi Y, Lee S. The Mediating Role of Sleep Disturbance on the Association Between Stress and Self-Rated Health Among Chinese and Korean Immigrant Americans. Prev Chronic Dis. 2023 Jan 26;20:E04. doi: 10.5888/pcd20.220241. PMID 36701271
- [Derived] Lee S, Ryu S, Lee GE, Redline S, Morey BN. Risk of Sleep Apnea Is Associated with Abdominal Obesity Among Asian Americans: Comparing Waist-to-Hip Ratio and Body Mass Index. J Racial Ethn Health Disparities. 2024 Feb;11(1):157-167. doi: 10.1007/s40615-022-01507-z. Epub 2023 Jan 9. PMID 36622567
- [Derived] Morey BN, Ryu S, Shi Y, Park HW, Lee S. Acculturation and Cardiometabolic Abnormalities Among Chinese and Korean Americans. J Racial Ethn Health Disparities. 2023 Aug;10(4):1605-1615. doi: 10.1007/s40615-022-01347-x. Epub 2022 Jun 15. PMID 35705844
- [Derived] Lee S, Ryu S, Lee GE, Kawachi I, Morey BN, Slopen N. The association of acculturative stress with self-reported sleep disturbance and sleep duration among Asian Americans. Sleep. 2022 Apr 11;45(4):zsab298. doi: 10.1093/sleep/zsab298. PMID 34922392

DOCUMENTS (2):
  • Study Protocol (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/96/NCT03481296/Prot_003.pdf
  • Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT03481296/SAP_004.pdf